CLINICAL TRIAL: NCT04700579
Title: Pre- and Post-treatment Lung Microbiota, Metabolome and Immune Signatures at the Site of Disease in Patients With Active Pulmonary Tuberculosis
Acronym: TB-LUNG
Status: Recruiting | Type: Observational
Sponsor: University of Stellenbosch (Other)
Collaborators: New York University (Other)
Responsible Party: Principal Investigator, Grant Theron, Professor, University of Stellenbosch
Other Study IDs: N19/09/126
Record Dates: First submitted 2020-12-28; First posted 2021-01-08 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: TB - Tuberculosis; HIV/AIDS
Keywords: Microbiome; Short Chain Fatty Acids; Immunological Biomarkers
MeSH Terms: conditions — Latent Tuberculosis; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — Bronchoalveolar lavage fluid, Protected specimen brushings, Sputum, Oro- Nasopharyngeal swabs, Urine, Blood and Stool.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- TB Cases: * n= 50 (25 HIV positive and 25 HIV negative)
  * Xpert MTB/RIF Ultra-confirmed TB
- Healthy Household Contacts: * n= (25 HIV positive and 25 HIV negative)
  * Culture negative TB result
- Sick controls: * n=50
  * Diseases: Asthma, Chronic obstructive pulmonary disease (COPD), Cancer, Bronchiectasis (including post-TB) and Pneumonia

SUMMARY:
The diverse microbial communities in different parts of the human body (microbiome) are important for health but understudied in pulmonary tuberculosis (TB), which is the single biggest infectious cause of death in the world. The investigators will study the site-of-disease microbiome (in the lung bronchoalveolar space) in TB cases to investigate how, before TB treatment, metabolic compounds made by microbes affect host biomarkers important for TB control. The investigators will ask this question again at the end-of-treatment and one year later. Specifically, the investigators will sample the lung at the active TB hotspot identified by imaging and compare this to a non-involved lung segment usually in the opposite lung. The investigators will compare the lung microbiome to other sites in the body (i.e. oral cavity, nasopharynx, supraglottis, and gut). A small amount of blood (~15 ml) will be collected to assess peripheral immunological correlates of the host microbiome. Protected specimen brushings of the lung will be used to explore transcriptomic signatures and how these relate to the lung microbiome. The investigators will also apply these questions to the same number of controls (healthy patients and patients with an alternative diagnoses). This will lay the foundation for clinical trials to evaluate if specific bacteria have diagnostic (e.g., PCR) or therapeutic potential (e.g., antibiotics, prebiotics, probiotics, vaccines) where targeting the microbiome could improve clinical outcomes.

DETAILED DESCRIPTION:
The human body is host to complex microbial communities at different anatomical sites such as the gut, oral cavity, vagina, skin, and the lower respiratory tract - a site previously thought to be sterile. Growing evidence has implicated the role of the human microbiome in various diseases for example, Prevotella-enriched lung communities in HIV-positive pneumonia patients independently predict 70-day mortality, and Lactobacillus enriched murine gut microbiome alleviates asthma-like symptoms. However, despite the scale and severity of TB, there are limited studies on the microbiome in TB cases, the site of disease, and the effect of treatment, especially in the context of HIV. These key knowledge gaps preclude the design and evaluation of interventions that could target the microbiome and avert poor treatment outcomes in TB.

To date the few microbiome studies in TB have focused on the upper respiratory tract (using specimens such as sputum) and gut rather than the site of disease which, in TB, is typically the lung. These studies have shown associations between the microbiome and state of disease. For example, mice colonized with Helicobacter hepaticus in the gut demonstrate poor control of mycobacterial growth, heightened inflammation, and severe tissue pathology in the lungs. The lung which is the site of disease in pulmonary TB has been widely considered sterile until recently and the lung microbiome remains widely understudied in TB regardless of the potential impact it might have in TB pathogenesis. One of the major reasons why the lung is understudied is the difficult in sampling the lung. The investigators will implement a modified bronchoscopy procedure to avoid microbial cross-contamination from neighbouring anatomical sites (including from diseased to healthy parts of the lungs) and to accurately sample the low biomass in the bronchoalveolar space. The investigators hypothesize that TB cases have a distinct site-of-disease lung microbiota compared to non-diseased contralateral tissue, characterized by an enrichment of oral anaerobic fermenters, SCFAs, and impaired inflammation and tissue repair biomarkers. They also expect microbial and host biomarkers to be altered by TB treatment. A study by one of the investigators has already demonstrated lung microbiomes enriched with anaerobic oral taxa are associated with lung inflammation of the Th17 phenotype. The products of microbial anaerobic metabolism have also been shown to modulate immune response to diseases. The investigators will correlate the complex microbial communities at the site-of-disease in TB with the microbial and host biomarkers at the site-of-disease.

The study will recruit self-reporting patients with their first TB episode and Xpert MTB/RIF Ultra-confirmed TB from Scottsdene and Wallacedene primary care clinics in Cape Town. A total of 50 TB cases equally stratified by HIV status and 50 healthy household contacts (HHC) also stratified by HIV will be recruited. In addition to HIV-negatives, the study is recruiting an equal number of ART-treated HIV-positive TB cases, because there an epidemiologically important subpopulation with impaired pulmonary immunity. An additional 50 sick controls with other pulmonary diseases (Asthma, Chronic obstructive pulmonary disease (COPD), Cancer, Bronchiectasis (including post-TB) and Pneumonia) will recruited as comparator groups.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old.
* Agree to undergo CXR and/or CT scan.
* Has unilateral TB disease defined as one lung with extensive evidence of TB disease (non-applicable to healthy controls; sick controls will require an alternative diagnosis).
* No evidence of prior TB treatment and/or CXR/CT does not have obvious evidence of prior TB.
* Willing to undergo a research bronchoscopy at baseline, 6 months and 18 months and likely to remain in the area for the study period.
* If HIV-positive, must be stable on antiretroviral therapy (ART) for ≥1 year.
* Able and willing to return for follow-up visits, with no plans to move in the near future.
* Willing to comply with study requirements i.e. provision of contact details and written, informed consent prior to enrolment.

Exclusion Criteria:

* Less than 18 years or older than 60 years of age.
* Has already initiated TB treatment.
* Rifampicin resistant.
* Has a previous history of TB.
* Bilateral TB disease defined as both lungs with extensive TB disease
* Has received probiotics, antibiotics or inhaled steroids within three months prior to enrolment (not applicable to sick controls)
* Has diabetes mellitus, which affects TB disease, treatment response, and the microbiome
* Has a contraindication for bronchoscopy (e.g., FEV1 <70%), as determined by bronchoscopists according to best practice guidelines
* Has a daily alcohol intake of more than 6 beers or 4 mixed drinks
* Is pregnant (a commercial human chorionic gonadotropin determination assay will be performed in accordance with manufacturer's guidance on urine) or pregnancy planned for follow-up period
* Recent hospitalization for any reason

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Self-presenting patients with Xpert MTB/RIF Ultra-confirmed TB (n=50, equally stratified by HIV) and culture negative HHCs (n=50, equally stratified by HIV) will be recruited from primary care clinics (Scottsdene and Wallacedene) in Cape Town, South Africa. An additional 50 sick controls with other lung diseases will be referred from Tygerberg Academic Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Characterization of changes in microbiota in diseased vs. non-diseased lung segments, stratified by HIV status. | Up to 18 months
  Lung microbiome in diseased and non-diseased segments determined by 16S rRNA gene sequencing.
Association of specific microbial taxa in diseased segments with elevated SCFAs and impaired host inflammation and tissue repair biomarkers. | Up to 18 months
  Correlation analysis of specific cytokines profiled using commercial multiplexed Luminex panels and SCFAs measured using Gas chromatography-mass spectrometry (GC-MS) assays.
Evaluate the impact of treatment on the lung microbiome. | Up to 18 months
  Characterize bacterial community resilience alongside changes in microbial and host biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Grant Theron, PhD, Principal Investigator — University of Stellenbosch
Locations (3):
- South Africa (3):
  - Kraaifontein Community Health Centre, Cape Town, Western Cape
  - Scottsdene Clinic, Cape Town, Western Cape
  - Wallacedene Clinic, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
Collaborators will have access to de-identified IPD data. Other researchers wishing to access the data will be required to sign a data sharing agreement as per institutional policies.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available once the findings are published.
Access Criteria: Data access will be granted to interested collaborators and parties through sharing of data files or login information for the study's secure RedCap electronic database during the course of patient recruitment.

REFERENCES:
- [Background] Yatsunenko T, Rey FE, Manary MJ, Trehan I, Dominguez-Bello MG, Contreras M, Magris M, Hidalgo G, Baldassano RN, Anokhin AP, Heath AC, Warner B, Reeder J, Kuczynski J, Caporaso JG, Lozupone CA, Lauber C, Clemente JC, Knights D, Knight R, Gordon JI. Human gut microbiome viewed across age and geography. Nature. 2012 May 9;486(7402):222-7. doi: 10.1038/nature11053. PMID 22699611
- [Background] Wade WG. The oral microbiome in health and disease. Pharmacol Res. 2013 Mar;69(1):137-43. doi: 10.1016/j.phrs.2012.11.006. Epub 2012 Nov 28. PMID 23201354
- [Background] Weiner J 3rd, Parida SK, Maertzdorf J, Black GF, Repsilber D, Telaar A, Mohney RP, Arndt-Sullivan C, Ganoza CA, Fae KC, Walzl G, Kaufmann SH. Biomarkers of inflammation, immunosuppression and stress with active disease are revealed by metabolomic profiling of tuberculosis patients. PLoS One. 2012;7(7):e40221. doi: 10.1371/journal.pone.0040221. Epub 2012 Jul 23. PMID 22844400
- [Background] Grice EA, Kong HH, Renaud G, Young AC; NISC Comparative Sequencing Program; Bouffard GG, Blakesley RW, Wolfsberg TG, Turner ML, Segre JA. A diversity profile of the human skin microbiota. Genome Res. 2008 Jul;18(7):1043-50. doi: 10.1101/gr.075549.107. Epub 2008 May 23. PMID 18502944
- [Background] Shenoy MK, Iwai S, Lin DL, Worodria W, Ayakaka I, Byanyima P, Kaswabuli S, Fong S, Stone S, Chang E, Davis JL, Faruqi AA, Segal MR, Huang L, Lynch SV. Immune Response and Mortality Risk Relate to Distinct Lung Microbiomes in Patients with HIV and Pneumonia. Am J Respir Crit Care Med. 2017 Jan 1;195(1):104-114. doi: 10.1164/rccm.201603-0523OC. PMID 27447987
- [Background] Wipperman MF, Fitzgerald DW, Juste MAJ, Taur Y, Namasivayam S, Sher A, Bean JM, Bucci V, Glickman MS. Antibiotic treatment for Tuberculosis induces a profound dysbiosis of the microbiome that persists long after therapy is completed. Sci Rep. 2017 Sep 7;7(1):10767. doi: 10.1038/s41598-017-10346-6. PMID 28883399
- [Background] Botero LE, Delgado-Serrano L, Cepeda ML, Bustos JR, Anzola JM, Del Portillo P, Robledo J, Zambrano MM. Respiratory tract clinical sample selection for microbiota analysis in patients with pulmonary tuberculosis. Microbiome. 2014 Aug 25;2:29. doi: 10.1186/2049-2618-2-29. eCollection 2014. PMID 25225609
- [Background] Cheung MK, Lam WY, Fung WY, Law PT, Au CH, Nong W, Kam KM, Kwan HS, Tsui SK. Sputum microbiota in tuberculosis as revealed by 16S rRNA pyrosequencing. PLoS One. 2013;8(1):e54574. doi: 10.1371/journal.pone.0054574. Epub 2013 Jan 24. PMID 23365674
- [Background] Cui Z, Zhou Y, Li H, Zhang Y, Zhang S, Tang S, Guo X. Complex sputum microbial composition in patients with pulmonary tuberculosis. BMC Microbiol. 2012 Nov 23;12:276. doi: 10.1186/1471-2180-12-276. PMID 23176186
- [Background] Segal LN, Clemente JC, Tsay JC, Koralov SB, Keller BC, Wu BG, Li Y, Shen N, Ghedin E, Morris A, Diaz P, Huang L, Wikoff WR, Ubeda C, Artacho A, Rom WN, Sterman DH, Collman RG, Blaser MJ, Weiden MD. Enrichment of the lung microbiome with oral taxa is associated with lung inflammation of a Th17 phenotype. Nat Microbiol. 2016 Apr 4;1:16031. doi: 10.1038/nmicrobiol.2016.31. PMID 27572644
- [Background] Segal LN, Alekseyenko AV, Clemente JC, Kulkarni R, Wu B, Gao Z, Chen H, Berger KI, Goldring RM, Rom WN, Blaser MJ, Weiden MD. Enrichment of lung microbiome with supraglottic taxa is associated with increased pulmonary inflammation. Microbiome. 2013 Jul 1;1(1):19. doi: 10.1186/2049-2618-1-19. PMID 24450871
- [Background] Naidoo CC, Nyawo GR, Wu BG, Walzl G, Warren RM, Segal LN, Theron G. The microbiome and tuberculosis: state of the art, potential applications, and defining the clinical research agenda. Lancet Respir Med. 2019 Oct;7(10):892-906. doi: 10.1016/S2213-2600(18)30501-0. Epub 2019 Mar 22. PMID 30910543